CLINICAL TRIAL: NCT03304028
Title: Use of Home-based Connected Devices to Early Detect and Treat Pulmonary Exacerbations: Feasibility and Clinical Validity in CF Patients
Brief Title: MUCOviscidose EXacerbation Outils Connectés Education Thérapeutique
Acronym: MucoExocet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment and search completed
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Fondation pour la Recherche Médicale (Other); Vertex Pharmaceuticals Incorporated (Industry); Fondation Ildys (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C16-119; 2017-A00723-50 (Registry Identifier: RCB)
Record Dates: First submitted 2017-09-22; First posted 2017-10-06 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Cystic Fibrosis
Keywords: Connected Devices; Pulmonary Exacerbations; Cumulative Sum (CUSUM) Chart
MeSH Terms: conditions — Cystic Fibrosis | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, longitudinal pilot study on cohort, in 3 phases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refusal Group (Other): Refusal Questionnaires Intervention:
  Clinic staff will email all patients or parents (pediatric settings) to introduce the study. A qualitative interview with 10 patients who declined to participate in the study will be conducted to identify the reason of refusal.
  Interventions: Behavioral: Refusal Questionnaires
- Interventionnal Group (Other): Connected Devices for 3 months (36 patients will be equipped with CDs-spirometer, oxymeter, scales, podometer watch and AURA device for sleep quality and analyze) Educationnal Intervention Connected Devices for 12 months Interviews
  Interventions: Device: Connected Devices for 3 months; Behavioral: Educationnal Intervention; Device: Connected Devices for 12 months; Other: Interviews

INTERVENTIONS:
Device: Connected Devices for 3 months — Inclusion will be proposed at a follow-up visit by the child's or adult's referring doctor. A written informed consent form will be obtained. Quality of Life and Anxiety-Depression will be collected. Then, each included patient will be equipped with CDs-spirometer, oxymeter, scale and watch during 3 months for base-line.
  Arms: Interventionnal Group
Behavioral: Educationnal Intervention — After a first statistical analysis and interpretation (5 months), alert parameters for each patient are then fixed. An educational visit will be scheduled with patients and a personnalized action plan will be defined..
  Arms: Interventionnal Group
Device: Connected Devices for 12 months — Each included patient will be re-equipped with CDs-spirometer, oxymeter, scale and watch during 12 months. If alerts occur, patients will be informed by email or SMS, with data transmission to the medical team who will not interfere. Patients should apply the shared action plan they learned. Quality of Life and Anxiety-Depression will be collected.
  Arms: Interventionnal Group
Other: Interviews — At the end, semi-structured interviews will be completed to explore confidence on the CDs, impact on the doctor-patient relationship, change in the workload of medical team…etc.
  Arms: Interventionnal Group
Behavioral: Refusal Questionnaires — Clinic staff will email all patients or parents (pediatric settings) to introduce the study. A qualitative interview with 10 patients who declined to participate in the study will be conducted to identify the reason of refusal
  Arms: Refusal Group

SUMMARY:
Early detection of pulmonary exacerbations (PEx) in Cystic Fibrosis (CF) patients is important to quickly trigger treatment and reduce respiratory damage. The investigators hypothesize that using home-based connected devices (CDs) in educated patients applying Cumulative sum charts (CUSUM) to monitor physiological parameters (PP) and patients' perception reported (PRP), will allow early detection of PEx.

Objective: to study clinical validity of using CDs and evaluate adherence and satisfaction in CF patients and teams

Design: 3 phase multicenter study in 36 CF patients aged >=12 years. Phase 1, patients are equipped during 3 months with CDs. PP and PRP to estimate CUSUM parameters are collected. In phase 2, patient's personalized educational plan to manage alerts is built. In phase 3, PP and PRP are collected during 12 months. Clinical validity, change in patients clinical data, quality of Life/Anxiety-Depression/Satisfaction, patients and teams' acceptance and adherence are assessed.

DETAILED DESCRIPTION:
BACKGROUND

Pulmonary exacerbations (PEx) are the major cause of lung function decline in Cystic Fibrosis (CF) patients leading to respiratory failure. Identifying warning signs of PEx is a priority to trigger early treatment and reduce respiratory damage. Some authors tried to define scores based on symptoms to standardize treatment. However, lack of consensus led the Euro-Care-CF-Working-Group to recommend the use of medical antibiotic treatment decision (or treatment modification) associated with PEx-like symptoms as best definition of PEx for clinical trials.

A DELPHI study identified 10 signs frequently perceived by patients and 10 most often cited indicators by caregivers. Two studies have shown that a combination of physiological parameters (PP) and patient reported perceptions (PRP) such as weight loss, decreased spirometry , increased cough or increased sputum production reported daily, help diagnose PEx episodes and trigger early treatment. Clinical observations show that changes in PP and PRP related to PEx differ according to age and degree of lung function impairment. Currently, patients with CF do not routinely monitor their lung function at home, nor do they objectively track PP or PRP. Consequently, CF PEx can be diagnosed late when symptoms progress, in which they seek medical care. Thus, development of an effective approach that helps to monitor daily indicators of PEx to early identification and treatment is important.

* Home monitoring of PEx symptoms Several studies have been conducted with daily monitoring of PEx symptoms. Most of these studies monitored one or two respiratory parameters with data transmission to the medical staff who decide what course of action to take. In addition, these studies used for each parameter the same alert limit for all patients, as it is known that patients with CF have different thresholds of these indicators,some may present more frequently than others.
* CUSUM to monitor indicators of pulmonary exacerbation The use of statistical process control (SPC) shows promise for monitoring indicators of CF PEx and rapidly detecting unwanted changes in these indicators. SPC uses rigorous time-series analysis methods, with results reported as a graph of changes in indicators over time[9]. Moreover, SPC can help to determine whether these changes are real (related to a causative factor) or merely a manifestation of natural variability. Among SPC, cumulative sum (CUSUM) chart has been found effective for measuring and monitoring healthcare outcome. It detects changes rapidly, and can identify small shifts. Connected devices software programming integrating CUSUM alert limits can help to determine whether the changes in PP and PRT are due to real PEx episode.

STUDY HYPOTHESIS The investigators hypothesize that using home-based CDs applying CUSUM with patient's personalized alert limits to monitor physiological data and PRP combined with patient education allows early detection of PEx. Studying alerts can help clinicians to develop a patient's personalized educational plan allowing patients better management of PEx including ability to make informed choices. This study aims to assess clinical validity of using different CDs, acceptance and adherence of patients of data collection of physiological data and PRPs, and acceptance by the clinical teams of this process of care. It will lead a larger trial aiming to evaluate efficacy of this process of care on patient's clinical outcomes.

DESIGN

Design: A 3 phase multi-center prospective longitudinal pilot study will be conducted.

- Phase 1- Baseline data collection Clinic staff will email all patients or parents (pediatric settings) to introduce the study. A qualitative interview with 10 patients who declined to participate in the study will be conducted to identify the reason of refusal.

M0: Inclusion visit: the inclusion will be proposed at a follow-up visit by the child's or adult's referring doctor. A written informed consent form will be obtained from all adults or both parents of children.

Quality of Life and Anxiety-Depression will be collected using the HADS and CFQ-R scale Each included patient will be equipped with CDs-spirometer, oxymeter, scale and watch During 3 months: Baseline data of 14 warning indicators of Pex will be collected during 3 non consecutive days a week using the CDs.

Number and time of acute PEx, FEV1, weight, respiratory symptoms and antibiotic treatments prescribed will be collected at the end of the period from the medical patient chart in the CF centre.

* Phase 2- statistical analysis and patient education Statistical analysis of the data collected in phase 1 will take place to calculate the CUSUM parameters. Alert parameters for each patient are then fixed. An educational visit will be scheduled with patients
* Phase 3- CDs use and personalized care PP and PRP will be continuously collected during 12 months using CDs. If alerts occur, patients will be informed by email or SMS, with data transmission to the medical team who will not interfere. Patients should apply the shared action plan they learned. Quality of Life and Anxiety-Depression will be collected using the HADS and CFQ-R scale. Number and time of acute PEx, FEV1, weight, respiratory symptoms and antibiotic treatments prescribed during the period will be collected at the end of the period from the medical patient chart in the CF centre.

At the end of Phase 3: Semi-structured interviews will be completed with the 30 patients/parents and 5 medical teams to explore confidence on the CDs, impact on the doctor-patient relationship, change in the workload of medical team…etc.

EXPECTED RESULTS

The investigators expect a better quality of life for patients, and that their anxiety-depression has not increased or rather decreased. For the clinical teams, the investigators aim to demonstrate that the use of CDs at home by educated patients is acceptable in their daily workload, and satisfying regarding the application of the shared action plan by the patient. Unlike other studies, patients are empowered to initiate actions when alerted by variations of the parameters. If they don't follow the action plan decided with the clinical teams, the treatment of PEx might not be earlier than if they didn't use CDs. In that case, a discussion with the clinicians may lead to the alternative process in which the alerts are used by the clinical teams to drive the actions for the patient. Interestingly, this alternative is possible because the alerts are simultaneously transmitted to the patient and to the team. The leader in the process may even change at some critical periods when the patient is in bad condition or depressed.

Qualitative analysis will provide knowledge on benefits and pitfalls to improve confidence in the use of CDS at home from the patients and the clinical teams, improve the patient-team partnership and, decrease stress and anxiety about pulmonary exacerbation treatment. This study will lead to further plan a larger trial aiming to evaluate efficacy of this process of care on patients' clinical outcomes

Scientific innovation The use of home based CD is rapidly growing and their contribution to the diagnosis of Pex in CF patients deserves to be fully evaluated. The use of CUSUM is particularly promising for monitoring indicators of CF PEx. Because CUSUM chart detects rapidly changes in these indicators and can identify small persistent shifts, it can help to trigger early treatment and reduce respiratory damages.

Furthermore, this is the first study which uses a combination of numerous CDs to evaluate several warning indicators of PEx. In addition, putting patients at the center of their health care and giving them more autonomy (empowerment) is innovative in this type of study and can improve both detection and management of their PEx episodes.

ELIGIBILITY:
Inclusion Criteria:

* 12 years and over
* Cystic fibrosis confirmed by sweat test or genetic
* Able to understand and respect the protocol and its requirements
* Who signed the consent prior to any other procedure protocolFollowed in the same CF center during the study
* In clinically stable condition - no pulmonary exacerbation requiring intravenous antibiotics - in the previous 4 weeks)
* Prescribed at least one pulmonary medication (eg, inhaled mucolytic, inhaled or oral antibiotic therapy, hypertonic saline)
* Not undergone solid organ transplants
* With smartphone, computer or tablet connected to wifi access

Exclusion Criteria:

* Patient undergoing solid organ transplant
* Pregnancy or planned pregnancy during the period of the study
* Patient on exclusion period because of other clinical research esearch
* Patients who don't use connected devices during the 3 first months will be excluded from the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Exacerbations (ExR) concordance | 2 Years
  Assesses agreement between the ExR episodes detected by the connected objects and the ExR episodes detected by the start date of the antibiotic treatment noted in the patient's medical record

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale (HADS) | Inclusion ; month 3 ; month 10 ; month 22
  Assesses anxiety and depressive disorders
Cystic Fibrosis Questionnaire-Revised (CFQ-R) | Inclusion ; month 3 ; month 10 ; month 22
  Assesses quality of live related to cystic fibrosis
Medical data : FEV1 | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses FEV1 (%) during a routine visit at the CF center
Medical data: Weight | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses weight (kilograms) during a routine visit at the CF center
Medical data: Height | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses height (meters) during a routine visit at the CF center
Medical data: Heart rate | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses heart rate during a routine visit at the CF center
Medical data: Oxygen saturation | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses oxygen saturation during a routine visit at the CF center
Physiological parameters with connected devices (PP) : FEV1 | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses with connected devices of FEV1 (%)
Physiological parameters with connected devices (PP) : Heart rate | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses with connected devices of heart rate
Physiological parameters with connected devices (PP) : Oxygen saturation | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses with connected devices of oxygen saturation
Physiological parameters with connected devices (PP) : Weight | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses with connected devices of weight (kilograms)
Physiological parameters with connected devices (PP) : Duration of sleep | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses with connected devices of duration of sleep
Physiological parameters with connected devices (PP) : Physical activity | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses with connected devices of physical activity (steps number)
Perceptions identified by patients (PRP) | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses by 1 questionnaire on connected devices of several illness perceptions (breathing difficulty ; need to intensify the physiotherapist ; increase in symptoms at night ; more sputum production ; increase in difficulty in daily activities ; tiredness ; reduction of appetite)
Traitements Number | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses number of antibiotic treatments prescribed during the study, collected from the data available in patient medical records
Traitements Duration | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses duration of antibiotic treatments prescribed during the study, collected from the data available in patient medical records
Respiratory symptoms | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses respiratory symptoms arising during the study, collected from the data available in patient medical records
Exacerbations Number | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses number acute exacerbations arising, collected from the data available in patient medical records
Exacerbations Timing | Inclusion ; month 3 ; month 10 ; month 13 ; month 16 ; month 19 ; month 22
  Assesses timing of acute exacerbations arising, collected from the data available in patient medical records
Patients and professionals interviews | 2 Years
  Assesses experiences and frequency of use of connected devices: factors influencing the use of connected devices, trust and conviction in connected devices, impact on physician-patient relationship, impact of connected devices on daily lives...
  Semi-structured interviews will be conducted
  * with the 30 patients: face to face or telephone
  * with the 7 participating medical teams: face to face

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RAULT, Ph, Principal Investigator — Fondation Ildys
Locations (7):
- France (7):
  - CF adults center - Hopital Albert Calmette, Lille
  - CF adults center - Institut du Thorax, Nantes
  - CF pediatrics center - Hopital Mère-Enfant, Nantes
  - CF pediatrics center - Hopital Robert Debré, Paris
  - CF adults and pediatrics center - American Memorial Hospital, Reims
  - CF adults and pediatrics center- Perharidy, Roscoff
  - CF pediatrics center - Hopital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Roux E, Ursino M, Milovanovic I, Picq P, Haignere J, Rault G, Pougheon Bertrand D, Alberti C. Home-Based Connected Devices Combined With Statistical Process Control for the Early Detection of Respiratory Exacerbations by Patients With Cystic Fibrosis: Pilot Interventional Study With a Pre-Post Design. JMIR Form Res. 2024 Oct 28;8:e51753. doi: 10.2196/51753. PMID 39467550
- [Derived] Morsa M, Perrin A, David V, Rault G, Le Roux E, Alberti C, Gagnayre R, Pougheon Bertrand D. Experiences Among Patients With Cystic Fibrosis in the MucoExocet Study of Using Connected Devices for the Management of Pulmonary Exacerbations: Grounded Theory Qualitative Research. JMIR Form Res. 2024 Jan 23;8:e38064. doi: 10.2196/38064. PMID 38261372
- [Derived] Morsa M, Perrin A, David V, Rault G, Le Roux E, Alberti C, Gagnayre R, Pougheon Bertrand D. Use of Home-Based Connected Devices in Patients With Cystic Fibrosis for the Early Detection and Treatment of Pulmonary Exacerbations: Protocol for a Qualitative Study. JMIR Res Protoc. 2021 Aug 18;10(8):e14552. doi: 10.2196/14552. PMID 34406124